CLINICAL TRIAL: NCT05023811
Title: A Phase I, Open-label Study of Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]RIST4721 Following a Single Oral Dose to Healthy Male Subjects
Brief Title: A Study of the ADME of [14C]RIST4721 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RIST4721-104
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Healthy; ADME

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [14C]RIST4721 (Experimental): [14C]RIST4721 oral solution
  Interventions: Drug: [14C]RIST4271

INTERVENTIONS:
Drug: [14C]RIST4271 — [14C]RIST4271 oral solution

SUMMARY:
A Phase I, Open-label Study of Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]RIST4721 Following a Single Oral Dose to Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Must provide written informed consent
* Body mass index (BMI) 18.0 to 30.0 kg/m2 as measured at screening
* Weight ≥50 kg and ≤100 kg inclusive at screening
* Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Evidence of current SARS-CoV-2 infection
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta: CumAe | Day 1 to Day 17
Mass balance recovery of total radioactivity in all excreta: Cum%Ae | Day 1 to Day 17
Determination of routes and rates of elimination of [14C]RIST4721 by Ae | Day 1 to Day 17
Determination of routes and rates of elimination of [14C]RIST4721 by %Ae | Day 1 to Day 17
Determination of routes and rates of elimination of [14C]RIST4721 by CumAe | Day 1 to Day 17
Determination of routes and rates of elimination of [14C]RIST4721 by Cum%Ae by interval | Day 1 to Day 17
Collection of plasma, urine and fecal samples for metabolite profiling | Day 1 to Day 17
Collection of plasma, urine and fecal samples for structural identification | Day 1 to Day 17
Collection of plasma, urine and fecal samples for quantification analysis | Day 1 to Day 17

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No